CLINICAL TRIAL: NCT03498196
Title: A Window of Opportunity Trial: Avelumab in Non-metastatic Muscle Invasive Bladder Cancer (BL-AIR: Bladder Cancer-Avelumab for Invasive Resectable Disease)
Brief Title: A Window of Opportunity Trial: Avelumab in Non-metastatic Muscle Invasive Bladder Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor of this study has terminated the study due to poor enrollment.
Sponsor: Baylor College of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jennifer Taylor, Assistant Professor of Urology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-41207
Record Dates: First submitted 2018-04-07; First posted 2018-04-13 (Actual); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Bladder Cancer; Metastatic Bladder Cancer; Invasive Bladder Cancer
Keywords: muscle invasive bladder cancer; non-muscle invasive bladder cancer; radical cystectomy; monoclonal antibodies; Avelumab; Invasive Resectable disease; MIBC; NMIBC; neoadjuvant chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental): Avelumab 10 mg/kg intravenously, over 60 minutes every 2 weeks for 3 cycles or 42 days.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — avelumab 10 mg/kg intravenously every 2 weeks for 3 cycles or 42 days.
  Other Names: MSB0010718C

SUMMARY:
This is a pilot study of avelumab in patients with non-metastatic, muscle invasive bladder cancer who are eligible for radical cystectomy (RC), but are ineligible for cisplatin based neoadjuvant therapy. The target recruitment is 10 evaluable patients for this window of opportunity study. Pre- and post-treatment tumor samples from transurethral resection of the bladder tumor and RC will be used for study endpoints.

DETAILED DESCRIPTION:
Avelumab is a fully human monoclonal PD-L1 antibody of the immunoglobulin G1 (IgG1) subclass. It works by binding to PD-L1 on tumor cells, immune cells and/or stromal cells. This prevents PD-L1 from interacting with PD-1. Inhibition of this interaction increases activation/survival of antitumor lymphocytes. It also increases innate immunity by resulting in decreased PD-1 suppression of NK cell function and bolsters antibody production by B cells due to less PD-L1 binding of PD-1 on B-cells. Additionally, avelumab has been suggested to have another mechanism involving antibody dependent cellular cytotoxicity (ADCC). ADCC in these cases involves NK cell recognition and lysis of tumor cells that have antibody bound to PD-L1. By blocking PD-L1, avelumab leads to less CD80 binding by PD-L1 and more CD80-CD28 binding in response to antigen presentation to T-cells. This results in increased costimulatory signaling and is another mechanism by which avelumab may enhance T-cell activation.

Avelumab has been shown to be efficacious across multiple metastatic tumor types, including urothelial cancer. The phase Ib study has reported survival and safety outcomes with >12 months followup using pooled data on 249 patients with metastatic UC (Apolo et al, ESMO Sept 2017). Patients had been treated with a median of 2 prior therapies in the metastatic setting and 13 patients who were cisplatin-ineligible were evaluated for safety alone. PD-L1 expression was not a criterion for enrollment. The confirmed objective response rate (ORR) was 16.1%, with 5% complete responses and 11.2% partial responses. The 6-month progression-free survival was 27%. The ORR was better than or comparable to chemotherapy in historical controls. Among responders, 70.3% were maintained > 12 months. Treatment-related adverse events (AE) occurred in 70%, with 10.7% of the total with AE's of grade >3. Immune-mediated AE's occurred in 18.5%, of which 4% were grade >3. There is currently a phase III clinical trial ongoing comparing avelumab to standard of care chemotherapy in the second line setting or beyond for metastatic UC. Two other checkpoint inhibitors have been approved in the last 2 years for first line treatment of patients with metastatic UC who are ineligible for cisplatin-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone TURBT showing newly diagnosed muscle invasive UCB (mixed histology is allowed if the predominant histology is UCC) within 6 weeks prior to cycle 1, day 1 of treatment.
* No prior systemic treatment for muscle invasive UCB
* Clinical T2-T4a disease
* No evidence of clinically positive lymph nodes or distant metastasis on computed tomography (CT) scans of chest and CT or magnetic resonance imaging (MRI) studies of the abdomen/pelvis. Imaging must be within 90 days of registration.
* Male or female subjects aged ≥ 18 years old.
* Must have adequate kidney, liver, and bone marrow function within 30 days of registration, as follows:
* Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
* platelet count ≥ 100 × 109/L
* hemoglobin ≥ 9 g/dL (may have been transfused)
* Total bilirubin level ≤ 1.5 × ULN
* AST and ALT levels ≤ 2.5 × ULN
* Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula
* Negative serum or urine pregnancy test at screening for women of childbearing potential (WOCBP), within 30 days of registration.
* Both male and female subjects must agree to use highly effective contraception (see Section 6.1 Table 8) while receiving avelumab and for at least 60 days after last avelumab treatment if the risk of conception exists.

Female patients must agree to inform study coordinator or investigator immediately if they think they have become pregnant during the study.

* Must have FFPE tissue available from the TURBT, and patient must consent to the use of tissue specimens from TURBT and RC for the study.
* Patients must be ineligible for cisplatin-based NAC. Ineligibility criteria include: creatinine clearance < 60 ml/min by Cockcroft-Gault formula, CTCAE grade ≥ 2 hearing loss, CTCAE grade ≥ 2 neuropathy, and at discretion of medical oncologist.
* Must be eligible for RC in the opinion of the treating investigator, and willing to undergo this procedure.
* ECOG performance status (PS) score of 0-2
* Signed informed consent form.

Exclusion Criteria:

Patients must not have any of the following:

* IMMUNOSUPRESSANTS: Current use of immunosuppressive medication or within 4 weeks of C1D1, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* AUTOIMMUNE DISEASE: Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible. Patients with type I diabetes or hypo- or hyperthyroidism should be on stable doses of medications for participation.
* ORGAN TRANSPLANTATION: Prior organ transplantation including allogenic stem-cell transplantation.
* INFECTIONS: Active infection requiring systemic therapy.
* HIV/AIDS: Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
* HEPATITIS: Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
* VACCINATION: Vaccinate within 4 weeks of the first dose of avelumab and while on study drug is prohibited except for administration of inactivated vaccines
* HYPERSENSITIIVTY TO STUDY DRUG: Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)
* CARDIOVASCULAR DISEASE: Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Relapsed MIBC (all patients participating in the study should be newly diagnosed)
* Concomitant UCC outside the bladder (e.g., ureter, urethra or renal pelvis)
* Underlying immune disorder (e.g., combined variable immunodeficiency syndrome)
* Erythropoietin receptor agonists within 30 days prior to enrollment.
* G-CSF, GM-CSF or TPO mimetics during the study period or within 3 weeks prior to study enrollment
* Malignancies other than UCB within 5 years prior to Cycle 1, Day 1, with the exception of those with low risk of metastasis or death treated with expected curative outcome (such as, but not limited to, adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent and absence of PSA relapse, or ductal carcinoma in situ of the breast treated surgically with curative intent) or incidental prostate cancer (T1a, Gleason score ≤ 6 and PSA < 0.5 ng/ml)
* Prior immunotherapy with T-cell co-stimulation or checkpoint targeted agents (e.g., CTLA-4 inhibitors, anti-PD1 antibodies or anti-PD-L1 antibodies)
* Intravesical chemotherapy or biologic therapy within 6 weeks of Cycle 1, Day 1
* Current participation in another clinical trial for MIBC
* Nursing or pregnant woman
* Uncontrolled cystitis, significant bladder pain or spasms, or gross hematuria that in the opinion of the principal investigator will preclude study participation
* Major surgical procedures within 4 weeks of registration (other than for diagnosis) or anticipation that such a procedure will be needed during the study (other than RC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M. Taylor, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor College of Medicine Medical Center - McNair Campus, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Michael E. DeBakey Veteran Affairs Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fairey AS, Daneshmand S, Quinn D, Dorff T, Dorin R, Lieskovsky G, Schuckman A, Cai J, Miranda G, Skinner EC. Neoadjuvant chemotherapy with gemcitabine/cisplatin vs. methotrexate/vinblastine/doxorubicin/cisplatin for muscle-invasive urothelial carcinoma of the bladder: a retrospective analysis from the University of Southern California. Urol Oncol. 2013 Nov;31(8):1737-43. doi: 10.1016/j.urolonc.2012.07.005. Epub 2012 Nov 7. PMID 23141776
- [Background] Galsky MD, Pal SK, Chowdhury S, Harshman LC, Crabb SJ, Wong YN, Yu EY, Powles T, Moshier EL, Ladoire S, Hussain SA, Agarwal N, Vaishampayan UN, Recine F, Berthold D, Necchi A, Theodore C, Milowsky MI, Bellmunt J, Rosenberg JE; Retrospective International Study of Cancers of the Urothelial Tract (RISC) Investigators. Comparative effectiveness of gemcitabine plus cisplatin versus methotrexate, vinblastine, doxorubicin, plus cisplatin as neoadjuvant therapy for muscle-invasive bladder cancer. Cancer. 2015 Aug 1;121(15):2586-93. doi: 10.1002/cncr.29387. Epub 2015 Apr 14. PMID 25872978
- [Background] Grossman HB, Natale RB, Tangen CM, Speights VO, Vogelzang NJ, Trump DL, deVere White RW, Sarosdy MF, Wood DP Jr, Raghavan D, Crawford ED. Neoadjuvant chemotherapy plus cystectomy compared with cystectomy alone for locally advanced bladder cancer. N Engl J Med. 2003 Aug 28;349(9):859-66. doi: 10.1056/NEJMoa022148. PMID 12944571
- [Background] Herchenhorn D, Dienstmann R, Peixoto FA, de Campos FS, Santos VO, Moreira DM, Cardoso H, Small IA, Ferreira CG. Phase II trial of neoadjuvant gemcitabine and cisplatin in patients with resectable bladder carcinoma. Int Braz J Urol. 2007 Sep-Oct;33(5):630-8; discussion 638. doi: 10.1590/s1677-55382007000500004. PMID 17980060
- [Background] International Collaboration of Trialists; Medical Research Council Advanced Bladder Cancer Working Party (now the National Cancer Research Institute Bladder Cancer Clinical Studies Group); European Organisation for Research and Treatment of Cancer Genito-Urinary Tract Cancer Group; Australian Bladder Cancer Study Group; National Cancer Institute of Canada Clinical Trials Group; Finnbladder; Norwegian Bladder Cancer Study Group; Club Urologico Espanol de Tratamiento Oncologico Group; Griffiths G, Hall R, Sylvester R, Raghavan D, Parmar MK. International phase III trial assessing neoadjuvant cisplatin, methotrexate, and vinblastine chemotherapy for muscle-invasive bladder cancer: long-term results of the BA06 30894 trial. J Clin Oncol. 2011 Jun 1;29(16):2171-7. doi: 10.1200/JCO.2010.32.3139. Epub 2011 Apr 18. PMID 21502557
- [Background] Plimack ER, Hoffman-Censits JH, Viterbo R, Trabulsi EJ, Ross EA, Greenberg RE, Chen DY, Lallas CD, Wong YN, Lin J, Kutikov A, Dotan E, Brennan TA, Palma N, Dulaimi E, Mehrazin R, Boorjian SA, Kelly WK, Uzzo RG, Hudes GR. Accelerated methotrexate, vinblastine, doxorubicin, and cisplatin is safe, effective, and efficient neoadjuvant treatment for muscle-invasive bladder cancer: results of a multicenter phase II study with molecular correlates of response and toxicity. J Clin Oncol. 2014 Jun 20;32(18):1895-901. doi: 10.1200/JCO.2013.53.2465. Epub 2014 May 12. PMID 24821881
- [Background] van de Putte EE, Mertens LS, Meijer RP, van der Heijden MS, Bex A, van der Poel HG, Kerst JM, Bergman AM, Horenblas S, van Rhijn BW. Neoadjuvant induction dose-dense MVAC for muscle invasive bladder cancer: efficacy and safety compared with classic MVAC and gemcitabine/cisplatin. World J Urol. 2016 Feb;34(2):157-62. doi: 10.1007/s00345-015-1636-y. Epub 2015 Jul 17. PMID 26184106
- [Background] Winquist E, Kirchner TS, Segal R, Chin J, Lukka H; Genitourinary Cancer Disease Site Group, Cancer Care Ontario Program in Evidence-based Care Practice Guidelines Initiative. Neoadjuvant chemotherapy for transitional cell carcinoma of the bladder: a systematic review and meta-analysis. J Urol. 2004 Feb;171(2 Pt 1):561-9. doi: 10.1097/01.ju.0000090967.08622.33. PMID 14713760
- [Background] Yeshchina O, Badalato GM, Wosnitzer MS, Hruby G, RoyChoudhury A, Benson MC, Petrylak DP, McKiernan JM. Relative efficacy of perioperative gemcitabine and cisplatin versus methotrexate, vinblastine, adriamycin, and cisplatin in the management of locally advanced urothelial carcinoma of the bladder. Urology. 2012 Feb;79(2):384-90. doi: 10.1016/j.urology.2011.10.050. Epub 2011 Dec 22. PMID 22196406
- [Background] Yuh BE, Ruel N, Wilson TG, Vogelzang N, Pal SK. Pooled analysis of clinical outcomes with neoadjuvant cisplatin and gemcitabine chemotherapy for muscle invasive bladder cancer. J Urol. 2013 May;189(5):1682-6. doi: 10.1016/j.juro.2012.10.120. Epub 2012 Nov 1. PMID 23123547
- [Background] Advanced Bladder Cancer (ABC) Meta-analysis Collaboration. Neoadjuvant chemotherapy in invasive bladder cancer: update of a systematic review and meta-analysis of individual patient data advanced bladder cancer (ABC) meta-analysis collaboration. Eur Urol. 2005 Aug;48(2):202-5; discussion 205-6. doi: 10.1016/j.eururo.2005.04.006. Epub 2005 Apr 21. PMID 15939524
- [Background] Bellmunt J, Ribas A, Eres N, Albanell J, Almanza C, Bermejo B, Sole LA, Baselga J. Carboplatin-based versus cisplatin-based chemotherapy in the treatment of surgically incurable advanced bladder carcinoma. Cancer. 1997 Nov 15;80(10):1966-72. doi: 10.1002/(sici)1097-0142(19971115)80:103.0.co;2-w. PMID 9366300
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Wolchok JD, Weber JS, Maio M, Neyns B, Harmankaya K, Chin K, Cykowski L, de Pril V, Humphrey R, Lebbe C. Four-year survival rates for patients with metastatic melanoma who received ipilimumab in phase II clinical trials. Ann Oncol. 2013 Aug;24(8):2174-80. doi: 10.1093/annonc/mdt161. Epub 2013 May 10. PMID 23666915
- [Background] Liu J, Hamrouni A, Wolowiec D, Coiteux V, Kuliczkowski K, Hetuin D, Saudemont A, Quesnel B. Plasma cells from multiple myeloma patients express B7-H1 (PD-L1) and increase expression after stimulation with IFN-gamma and TLR ligands via a MyD88-, TRAF6-, and MEK-dependent pathway. Blood. 2007 Jul 1;110(1):296-304. doi: 10.1182/blood-2006-10-051482. Epub 2007 Mar 15. PMID 17363736
- [Background] Taube JM, Anders RA, Young GD, Xu H, Sharma R, McMiller TL, Chen S, Klein AP, Pardoll DM, Topalian SL, Chen L. Colocalization of inflammatory response with B7-h1 expression in human melanocytic lesions supports an adaptive resistance mechanism of immune escape. Sci Transl Med. 2012 Mar 28;4(127):127ra37. doi: 10.1126/scitranslmed.3003689. PMID 22461641
- [Background] Daud AI, Wolchok JD, Robert C, Hwu WJ, Weber JS, Ribas A, Hodi FS, Joshua AM, Kefford R, Hersey P, Joseph R, Gangadhar TC, Dronca R, Patnaik A, Zarour H, Roach C, Toland G, Lunceford JK, Li XN, Emancipator K, Dolled-Filhart M, Kang SP, Ebbinghaus S, Hamid O. Programmed Death-Ligand 1 Expression and Response to the Anti-Programmed Death 1 Antibody Pembrolizumab in Melanoma. J Clin Oncol. 2016 Dec;34(34):4102-4109. doi: 10.1200/JCO.2016.67.2477. Epub 2016 Oct 31. PMID 27863197
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Rosenberg JE, Hoffman-Censits J, Powles T, van der Heijden MS, Balar AV, Necchi A, Dawson N, O'Donnell PH, Balmanoukian A, Loriot Y, Srinivas S, Retz MM, Grivas P, Joseph RW, Galsky MD, Fleming MT, Petrylak DP, Perez-Gracia JL, Burris HA, Castellano D, Canil C, Bellmunt J, Bajorin D, Nickles D, Bourgon R, Frampton GM, Cui N, Mariathasan S, Abidoye O, Fine GD, Dreicer R. Atezolizumab in patients with locally advanced and metastatic urothelial carcinoma who have progressed following treatment with platinum-based chemotherapy: a single-arm, multicentre, phase 2 trial. Lancet. 2016 May 7;387(10031):1909-20. doi: 10.1016/S0140-6736(16)00561-4. Epub 2016 Mar 4. PMID 26952546
- [Background] Huang RY, Eppolito C, Lele S, Shrikant P, Matsuzaki J, Odunsi K. LAG3 and PD1 co-inhibitory molecules collaborate to limit CD8+ T cell signaling and dampen antitumor immunity in a murine ovarian cancer model. Oncotarget. 2015 Sep 29;6(29):27359-77. doi: 10.18632/oncotarget.4751. PMID 26318293
- [Background] Woo SR, Turnis ME, Goldberg MV, Bankoti J, Selby M, Nirschl CJ, Bettini ML, Gravano DM, Vogel P, Liu CL, Tangsombatvisit S, Grosso JF, Netto G, Smeltzer MP, Chaux A, Utz PJ, Workman CJ, Pardoll DM, Korman AJ, Drake CG, Vignali DA. Immune inhibitory molecules LAG-3 and PD-1 synergistically regulate T-cell function to promote tumoral immune escape. Cancer Res. 2012 Feb 15;72(4):917-27. doi: 10.1158/0008-5472.CAN-11-1620. Epub 2011 Dec 20. PMID 22186141
- [Background] Sweis RF, Spranger S, Bao R, Paner GP, Stadler WM, Steinberg G, Gajewski TF. Molecular Drivers of the Non-T-cell-Inflamed Tumor Microenvironment in Urothelial Bladder Cancer. Cancer Immunol Res. 2016 Jul;4(7):563-8. doi: 10.1158/2326-6066.CIR-15-0274. Epub 2016 May 17. PMID 27197067
- [Background] Carthon BC, Wolchok JD, Yuan J, Kamat A, Ng Tang DS, Sun J, Ku G, Troncoso P, Logothetis CJ, Allison JP, Sharma P. Preoperative CTLA-4 blockade: tolerability and immune monitoring in the setting of a presurgical clinical trial. Clin Cancer Res. 2010 May 15;16(10):2861-71. doi: 10.1158/1078-0432.CCR-10-0569. Epub 2010 May 11. PMID 20460488
- [Background] Massard C, Gordon MS, Sharma S, Rafii S, Wainberg ZA, Luke J, Curiel TJ, Colon-Otero G, Hamid O, Sanborn RE, O'Donnell PH, Drakaki A, Tan W, Kurland JF, Rebelatto MC, Jin X, Blake-Haskins JA, Gupta A, Segal NH. Safety and Efficacy of Durvalumab (MEDI4736), an Anti-Programmed Cell Death Ligand-1 Immune Checkpoint Inhibitor, in Patients With Advanced Urothelial Bladder Cancer. J Clin Oncol. 2016 Sep 10;34(26):3119-25. doi: 10.1200/JCO.2016.67.9761. Epub 2016 Jun 6. PMID 27269937
- [Background] Sharma P, Callahan MK, Bono P, Kim J, Spiliopoulou P, Calvo E, Pillai RN, Ott PA, de Braud F, Morse M, Le DT, Jaeger D, Chan E, Harbison C, Lin CS, Tschaika M, Azrilevich A, Rosenberg JE. Nivolumab monotherapy in recurrent metastatic urothelial carcinoma (CheckMate 032): a multicentre, open-label, two-stage, multi-arm, phase 1/2 trial. Lancet Oncol. 2016 Nov;17(11):1590-1598. doi: 10.1016/S1470-2045(16)30496-X. Epub 2016 Oct 9. PMID 27733243
- [Background] Bellmunt J, de Wit R, Vaughn DJ, Fradet Y, Lee JL, Fong L, Vogelzang NJ, Climent MA, Petrylak DP, Choueiri TK, Necchi A, Gerritsen W, Gurney H, Quinn DI, Culine S, Sternberg CN, Mai Y, Poehlein CH, Perini RF, Bajorin DF; KEYNOTE-045 Investigators. Pembrolizumab as Second-Line Therapy for Advanced Urothelial Carcinoma. N Engl J Med. 2017 Mar 16;376(11):1015-1026. doi: 10.1056/NEJMoa1613683. Epub 2017 Feb 17. PMID 28212060
- [Background] Balar AV, Galsky MD, Rosenberg JE, Powles T, Petrylak DP, Bellmunt J, Loriot Y, Necchi A, Hoffman-Censits J, Perez-Gracia JL, Dawson NA, van der Heijden MS, Dreicer R, Srinivas S, Retz MM, Joseph RW, Drakaki A, Vaishampayan UN, Sridhar SS, Quinn DI, Duran I, Shaffer DR, Eigl BJ, Grivas PD, Yu EY, Li S, Kadel EE 3rd, Boyd Z, Bourgon R, Hegde PS, Mariathasan S, Thastrom A, Abidoye OO, Fine GD, Bajorin DF; IMvigor210 Study Group. Atezolizumab as first-line treatment in cisplatin-ineligible patients with locally advanced and metastatic urothelial carcinoma: a single-arm, multicentre, phase 2 trial. Lancet. 2017 Jan 7;389(10064):67-76. doi: 10.1016/S0140-6736(16)32455-2. Epub 2016 Dec 8. PMID 27939400
- [Background] Oing C, Rink M, Oechsle K, Seidel C, von Amsberg G, Bokemeyer C. Second Line Chemotherapy for Advanced and Metastatic Urothelial Carcinoma: Vinflunine and Beyond-A Comprehensive Review of the Current Literature. J Urol. 2016 Feb;195(2):254-63. doi: 10.1016/j.juro.2015.06.115. Epub 2015 Sep 26. PMID 26410730
- See also: SITC 2016: Immune Checkpoint Inhibitors Shrink Tumors in Some Patients With Metastatic Bladder Cancer — http://www.ascopost.com/News/44121
- See also: Cardiac Complications in Patients Receiving Combination Checkpoint Inhibitors Are Rare but Can Be Fatal — http://www.ascopost.com/issues/december-10-2016/cardiac-complications-in-patients-receiving-combination-checkpoint-inhibitors-are-rare-but-can-be-fatal/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Avelumab
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avelumab
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (NA) — there is only one participant.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
Current Smoking [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in T Cell Subpopulations
Description: The change in T cell subpopulations (CD8, CD4 and/or CD3) in tumor samples will be collected from FFPE tissue. FFPE tissue from the pre-study time point refers to tissue from the TURBT. FFPE tissue from the 2-3 week post-op time point refers to FFPE tissue from the RC
Time Frame: pre-study time and 2-3 week post-operation
Population: The assay for the outcome measure was planned to do after enrolling several patients and collecting specimen but only one patient was enrolled for this study. No assay was done.
Arm/Group | Avelumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Pathological Response Rate
Description: Number of patient with pathological response will be counted
Time Frame: pre-study time and 2-3 week post-operation
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: 2 Year Disease Free Survival (DFS)
Description: A patient will be followed for recurrence and survival for up to 2 years after radical cystectomy.
Time Frame: 2 years after radical cystectomy
Population: since one patient was available for this study analysis, the time of recurrence or death was reported.
Measure: Number; unit: months
Arm/Group | Avelumab
Number analyzed (Participants) | 1
months | 5.48

4. Secondary Outcome: Rate of High Grade(Grade 3-4) Adverse Event
Description: High grade adverse events are defined as grade of 3-4 on the CTCAE (Common terminology criteria for adverse events) grading scale.
Time Frame: 90 days post operation
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 90 days after radical cystectomy (RC) or end of the last cycle of Avelumab for those not receiving RC.
Arm/Group | Avelumab
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab (N=1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (3)
Creatinine increased (Investigations) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT03498196/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT03498196/SAP_001.pdf